CLINICAL TRIAL: NCT03657017
Title: PET/MR in Locally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET/MR-2018-01
Record Dates: First submitted 2018-08-15; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Nasopharyngeal Carcinoma; PET/MR
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MR (Other): Patients are examined with PET/MR.
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — Performed on a hybrid PET/MR scanner before treatment start (N = 150). Among those patients, 10 patients are examined with PET/MR in the completion of neoadjuvant chemotherapy and a follow-up scan three months after the completion of radiotherapy.

SUMMARY:
PET/MR in Locally Advanced Nasopharyngeal Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing carcinoma.
* Tumor staged T1-4N0-3M0 （according to the 8th AJCC staging system）
* Performance status: KPS>70
* With normal liver function test (ALT, AST <1.5ULN)
* Renal: creatinine clearance >60ml/min
* Without hematopathy,marrow: WBC >4*109/L, HGB>80G/L, and PLT>100*109/L.
* Written informed consent

Exclusion Criteria:

* Adenocarcinoma
* Age >70
* Prior malignancy (except adequately treated carcinoma in-situ of the cervix or · basal/squamous cell carcinoma of the skin)
* Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume)
* Patient is pregnant or lactating
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), or emotional disturbance.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Multiparametric PET/MRI-based radiomics nomograms for locally advanced nasopharyngeal carcinoma | From day 1 of chemotherapy to the date of the event, a minimum follow-up of 3 years.
  Radiomics-based prognostic model by PET/MRI

SECONDARY OUTCOMES:
Prediction model of the efficiency of treatment in locally advanced nasopharyngeal carcinoma | about 4 years (all of patients complete treatment)
  Radiomics-based prediction model of the efficiency of treatment by PET/MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No